CLINICAL TRIAL: NCT06755294
Title: Vestibular Incision Subperiosteal Tunnel Access (VISTA) Technique Versus Coronally Advanced Flap (CAF) Combined With a Connective Tissue Graft for the Treatment of Maxillary Gingival Recessions: a Randomized Clinical Trial
Brief Title: Vestibular Incision Subperiosteal Tunnel Access (VISTA) Technique Versus Coronally Advanced Flap (CAF) Combined With a Connective Tissue Graft for the Treatment of Maxillary Gingival Recessions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Alvaro Babiano Nodal, DDS/MsC, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PER-ECL-2023-09
Record Dates: First submitted 2024-12-23; First posted 2025-01-01 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Gingival Recessions
Keywords: VISTA TECHNIQUE; CAF; Root Coverage
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEST (Experimental): VISTA TECHNIQUE
  Interventions: Procedure: Vestibular incision subperiostal tunnel technique
- Control (Experimental): Coronally Advanced Technique
  Interventions: Procedure: CAF

INTERVENTIONS:
Procedure: Vestibular incision subperiostal tunnel technique — The VISTA (Vestibular Incision Subperiosteal Tunnel Access) technique is a minimally invasive surgical approach for root coverage. A single vertical incision is made, often at the labial frenulum for optimal access, reaching the periosteum to elevate a subperiosteal tunnel. This tunnel is extended beyond the mucogingival junction and interproximally under each papilla to enable tension-free coronal repositioning of the gingiva.
  An autologous connective tissue graft, harvested and de-epithelialized from the palate, is introduced into the tunnel. Before placement, teeth are etched (orthophosphoric or hydrofluoric acid depending on surface type). Sutures (6-0 polypropylene) stabilize the graft, with additional composite fixation on treated teeth. The vertical incision is closed using 5-0 sutures, ensuring proper stabilization and healing. This approach minimizes trauma, promotes healing, and achieves effective root coverage.
  Arms: TEST
Procedure: CAF — The Coronally Advanced Flap (CAF) is an effective technique for root coverage in single or multiple gingival recession cases with adequate apical keratinized tissue thickness and height. Following the De Sanctis and Zucchelli protocol (2007), two horizontal incisions are made 3 mm apart, with placement 1 mm apical to the recession height. Vertical beveled incisions extend into the alveolar mucosa, and a flap is elevated in three stages: partial thickness at the papilla, full thickness to the buccal bone table, and apical partial thickness to release muscle fibers for mobility.
  An autologous connective tissue graft (≥1 mm thick) is harvested from the palatal or retromolar area, de-epithelialized, and shaped to the recession size. The anatomical papillae are de-epithelialized, and the graft is sutured apically to the CEJ using 6-0 Polyglactin 910. Sling sutures (6-0 polypropylene) stabilize the flap 2 mm coronally to the CEJ, ensuring optimal positioning and healing.
  Arms: Control

SUMMARY:
Gingival recession (GR) is a common oral health problem that causes sensitivity, esthetic concerns and hygiene problems. Successful root coverage can be achieved by various surgical techniques. The VISTA technique may overcome some of the limitations of other techniques and present equal results to techniques that are considered the "Gold Standard" in this area of periodontology.

The objective of the research is to study the VISTA technique in terms of complete root coverage, % root coverage, gingival thickness gain, bleeding on probing, keratinized gingival width, PROMS, vestibular depth and esthetic results.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults: men and women between 18 and 75 years of age.
* Accepts and signs informed consent.
* Systemically healthy patients with periodontal health or controlled periodontitis.
* Presence of at least two maxillary Cairo Type I or II (RT1/2) recessions > 2 mm deep on buccal aspect.
* Plaque index ≤20%
* No previous periodontal surgeries performed.
* Presence of the cementoenamel junction (CEJ), a 1 mm step in the CEJ and/or presence of root abrasion, but with an identifiable CEJ will be accepted.

Exclusion Criteria:

* Smoker of 10 ≥ cigarettes per day.
* Contraindications to periodontal surgery.
* Medications that affect the gingiva or their healing.
* Active orthodontic treatment.
* Pregnant women
* Caries or restorations in the area to be treated.
* Patients who cannot follow the post-surgical medication adequately

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Recession reduction (RR) | 3 months and 6 months after the surgery
  Measured with a periodontal probe and with a STL file

SECONDARY OUTCOMES:
mean root coverage (% RC) | 3 and 6 months after the surgery
  Measured with a periodontal probe and with a STL file
PPD | Baseline, 3 and 6 months after the surgery
  distance from the gingival margin to the base of the gingival sulcus
CAL | Baseline, 3 and 6 months after the surgery
  distance from the LAC to the base of the gingival sulcus
KTW | Baseline, 3 and 6 months after the surgery
  distance from the gingival margin to the mucogingival line (MGL
Gingival thickness | Baseline, 3 and 6 months after the surgery
  Distance from the most external part of the gingiva to the buccal plate. Measured with a periodontal probe and with a STL file
Complete root coverage | 3 and 6 months after the surgery
  Measured with a periodontal probe and with a STL file